CLINICAL TRIAL: NCT05939843
Title: Brief Mindfulness for Foot and Ankle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam Hanley, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB_00085446 2
Record Dates: First submitted 2023-06-26; First posted 2023-07-11 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Single Person

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pain Coping Information (Active Comparator)
  Interventions: Behavioral: Pain Coping Information
- Mindfulness Practice (alone) (Experimental)
  Interventions: Behavioral: Mindfulness Practice (alone)
- Mindfulness Introduction + Mindfulness Practice (Experimental)
  Interventions: Behavioral: Mindfulness Introduction + Mindfulness Practice
- Pain Introduction + Mindfulness Introduction + Mindfulness Practice (Experimental)
  Interventions: Behavioral: Pain Introduction + Mindfulness Introduction + Mindfulness Practice

INTERVENTIONS:
Behavioral: Pain Coping Information — A three minute audio recording providing common pain coping techniques (e.g., ice, rest, medication, surgery)
  Arms: Pain Coping Information
Behavioral: Mindfulness Practice (alone) — A 3-minute audio-guided mindfulness practice.
  Arms: Mindfulness Practice (alone)
Behavioral: Mindfulness Introduction + Mindfulness Practice — A 1-minute audio-recorded introduction to the practice of mindfulness followed by a 2-minute audio-guided mindfulness practice
  Arms: Mindfulness Introduction + Mindfulness Practice
Behavioral: Pain Introduction + Mindfulness Introduction + Mindfulness Practice — A 1-minute audio-recorded introduction to pain, followed by a 1-minute audio-recorded introduction the practice of mindfulness, followed by a 1-minute audio-guided mindfulness practice
  Arms: Pain Introduction + Mindfulness Introduction + Mindfulness Practice

SUMMARY:
This is a single-site, four-arm, parallel-group randomized clinical trial (RCT). The clinical effects of three different formats of a very brief (i.e., 3 minute), audio-recorded mindfulness intervention for foot and ankle patients will be investigated relative to a 3-minute audio-recoding about pain psychoeducation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Seeking foot or ankle treatment at the University Orthopaedic Center

Exclusion Criteria:

* Cognitive impairment preventing completion of study procedures.
* Current cancer diagnosis,
* Other unstable illness judged by medical staff to interfere with study involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Change in Pain Unpleasantness Numeric Rating Scale | Immediately before to after 3-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most unpleasant pain imaginable.

SECONDARY OUTCOMES:
Change in Pain Intensity Numeric Rating Scale | Immediately before to after 3-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no pain and 10 representing the most intense pain imaginable.
Change in Pain Medication Desire Numeric Rating Scale | Immediately before to after 3-minute audio recording
  Single Likert scale item ranging from 0-10, with 0 indicating no desire for pain medication and 10 representing a strong desire for pain medication.

OTHER OUTCOMES:
Postoperative Patient Reported Outcomes Measurement Information System (PROMIS) Physical Functioning Item Bank, v2.0 | From before the patient's intervention visit to their subsequent re-evaluation. This time span is typically around 6 weeks.
  The PROMIS physical functioning computer assisted test draws from a bank of 123 items all scored on a 5 point Likert scale.
  T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. A high score better physical functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States